CLINICAL TRIAL: NCT06518824
Title: Theta Deep Brain Stimulation for Cognitive Enhancement in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Stefan Lang, MD, PhD FRCSC, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: thetaDBS
Record Dates: First submitted 2024-07-10; First posted 2024-07-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Cognitive Impairment
Keywords: Theta Stimulation
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stimulation off (Sham Comparator): The deep brain stimulation device will be turned off.
  Interventions: Device: DBS Off
- Theta stimulation of associative STN region (Experimental): The deep brain stimulation device will be set to a frequency of 6 Hz and will stimulate the associative STN region. If differential activation of the associative and sensorimotor STN networks is not feasible, ventral stimulation is employed.
  Interventions: Device: DBS On
- Theta stimulation of STN sensorimotor region (Active Comparator): The deep brain stimulation device will be set to a frequency of 6 Hz and will stimulate the sensorimotor region, acting as an anatomical control. If differential activation of the associative and sensorimotor STN networks is not feasible, dorsal stimulation is employed.
  Interventions: Device: DBS On
- High frequency stimulation of associative STN region (Active Comparator): The deep brain stimulation device will be set to a frequency of 135 Hz and will stimulate the associative STN region, acting as a frequency control. If differential activation of the associative and sensorimotor STN networks is not feasible, ventral VTA is employed.
  Interventions: Device: DBS On

INTERVENTIONS:
Device: DBS On — The DBS device will be turned on while the patient undergoes the working memory task.
  Arms: High frequency stimulation of associative STN region; Theta stimulation of STN sensorimotor region; Theta stimulation of associative STN region
Device: DBS Off — The DBS device will be turned off while the patient undergoes the working memory task.
  Arms: Stimulation off

SUMMARY:
Cognitive impairment is common in Parkinson's disease. A recent study demonstrated 40% of people with PD suffer from mild cognitive impairment and > 80% of patients develop dementia after a disease duration of 20 years. Cognitive impairment significantly impairs quality of life and has limited treatment options. While the pathophysiology of cognitive symptoms in PD is multifactorial, one contributing factor is dysfunction in subthalamic-cortical loops.

The subthalamic nucleus (STN) receives input from distributed regions of the cortex, forming partially segregated parallel networks with sensorimotor regions, associative (cognitive) cortical regions, and limbic cortical regions. These subthalamic-cortical networks are thought to play a domain general role in inhibitory control, which is a fundamental mechanism underlying flexible behavior across motor, cognitive, and affective domains. Information processing in these subthalamic-cortical networks is expressed through oscillatory activity within distinct frequency bands. For example, communication between the STN and prefrontal regions involved in executive function is thought to occur through coherence in the theta (4-8 Hz) frequency band. As a result of these observations, stimulation of the STN at a theta frequency has been investigated as a method of modulating cognitive processes.

Theta stimulation of the STN has been shown to enhance coherence in subthalamic-cortical networks, facilitating information processing and modulating behavior. For example, a recent study demonstrated that theta stimulation of the STN improved working memory performance in PD subjects, while no effect was seen for other frequency bands. The authors performed a post-hoc analysis and found that the effect may be mediated by connectivity between the stimulated STN region and the right dorsolateral prefrontal cortex (DLPFC). While these studies have demonstrated proof of principle, they are limited by small sample sizes and post-hoc analyses assessing the relationship between stimulation location and outcomes. Further research is needed to directly test the hypothesis that theta stimulation of the STN can improve executive control in PD patients by modulating associative STN circuitry.

DETAILED DESCRIPTION:
Objective: The objective of the proposed research is to test the ability of theta stimulation of the STN to modulate cognitive processing in PD patients by directly targeting associative STN circuitry.

Hypothesis: The hypothesis is that theta stimulation of associative STN circuitry will improve performance on cognitive tasks compared to a control condition, where stimulation is targeting a sensorimotor STN circuit.

Methods: Power analysis - with previously reported moderate effect sizes (Cohen's d=0.57), the investigators anticipate the need to recruit 27 subjects for a within-subject design with a power of 0.8 and an alpha level of 0.05.

Subjects: Patients with deep brain stimulation systems will be recruited from the Vancouver General Hospital DBS clinic. Subjects will be included if they have STN DBS, pre- and post-operative imaging (to allow electrode reconstruction), and are at least three months post-operative. Subjects will be excluded if they are unable to complete the cognitive task (due to language barriers or dementia) or if they have significant DBS related complications.

Study design: This is a double blind, randomized, cross-over within-subject repeated measure design assessing the interaction between stimulation location and behavioural modification. Subjects will be blinded to stimulation condition, and the individual administering the working memory task will also be blinded, as a neutral third party will program the DBS settings for each condition.

Identification of associative STN network and optimal electrode configuration: Before the subject arrives for stimulation, the location of the electrode will be reconstructed using the pipeline in LeadDBS. Briefly, a pre-operative MRI and a post-operative CT scan will be co-registered and subsequently non-linearly normalized into standard space. Electrodes will be identified and reconstructed using the PaCER algorithm as implemented in LeadDBS. Using each subject's individualized electrode reconstruction, we will calculate the volume of tissue activated (VTA) to optimally engage either the associative or sensorimotor STN networks. Multiple VTA configurations will be evaluated to achieve this goal. VTAs targeting the associative STN network will be defined by maximizing structural and functional connectivity to the dorsolateral prefrontal cortex (DLPFC) while minimizing connectivity to the primary motor cortex (M1) and supplementary motor area (SMA) among the viable configurations for the individual electrode. Conversely, VTAs designed to engage the sensorimotor STN network are defined by maximizing connectivity to M1 and SMA and minimizing connectivity to the DLPFC.

Structural and functional connectivity will be quantified as follows: Percent overlap of the individual VTA with the associative and sensorimotor STN regions will be calculated using MATLAB, employing the DISTAL Atlas to delineate each STN region. Structural connectivity will be estimated by computing the total number of streamlines connected to the VTA that pass through the specified region-of-interest (ROI), based on structural normative connectomes. Functional connectivity will be assessed by calculating the Pearson's correlation coefficient between the VTA and the ROI, using resting-state functional normative connectomes.

If it is not feasible to differentially activate the associative or sensorimotor STN networks using these criteria, simplified VTAs will be employed: a ventral VTA and a dorsal VTA. This may be the case due to the anatomical location of the electrode or the electrode model (ring-mode or directional).

Baseline cognitive assessment: Each subject will undergo a baseline cognitive screening examination (Montreal Cognitive Assessment, MOCA), that will be used as a covariate in future analysis. This will be done as part of their routine screening prior to DBS surgery.

Theta DBS: Subjects will come into the clinic in the OFF-medication state, to help control for the known non-linear contribution of dopamine to working memory. They will undergo a computerized working memory task while being stimulated in each of four following conditions:

1. OFF
2. Target condition: Theta (6 Hz) stimulation of the associative STN. If differential activation of the associative and sensorimotor STN networks is not feasible, ventral VTA is used.
3. Anatomical control condition: Theta stimulation of the sensorimotor STN. If differential activation is not feasible, dorsal VTA is used
4. Frequency control condition: High-frequency (135 Hz) stimulation of the associative STN. If differential activation is not feasible, ventral VTA is used.

These conditions will be randomized within each subject by creating a random integer (1-4) with no repeats. The amplitude and pulse width will remain constant (2.5 mA, 60us). After changing the stimulation setting, there will be a wait period of 5-10 minutes prior to commencement of the working memory task. The subject will be asked if there is any unwanted stimulation side-effect (for example paresthesia). If the subject has paraesthesia or otherwise complains about the stimulation, the amplitude will be reduced by 0.5mA. If stimulation is not possible, the patient will be excluded from the study. Immediately before the working memory task commences, subjects will undergo a brief motor examination, consisting of items from the Unified Parkinson's Disease Rating Scale III. At the end of the session, the subjects will be placed back on their clinically optimized program and will take their medication according to their normal schedule.

Working Memory Task: A modified Sternberg task will be presented using a laptop computer.

Statistical analysis: The primary outcome will be working memory performance during each stimulation condition as assessed by a linear mixed effect model. The model will be specified as working memory performance ~ age + MoCA + stimulation condition + baseline cognition*stimulation condition + stimulation order + (1|subject). The hypothesis is that there will be a main effect of stimulation condition on working memory performance, with post-hoc one sample t-tests demonstrating an improvement in the theta associative STN condition relative to the other conditions. An interaction effect of baseline cognition with stimulation condition is also expected to be observed. Based on previous literature, it is hypothesized that subjects with lower baseline cognition will have more improvement during associative STN region stimulation.

To further understand the impact of differential network activation, a secondary analysis will categorize subjects into two groups: 1) those where differential activation of the associative and sensorimotor STN networks was achieved and 2) those where differential targeting of these networks was not possible based on the imaging criteria. We will repeat the linear mixed effect model, adding an interaction term between stimulation condition and group. The hypothesis is that there will be a significant interaction effect between stimulation condition and group, with higher working memory performance observed during theta stimulation of the associative STN in the group where differential targeting of the associative STN network was achieved. This will enable the assessment of whether precise STN network targeting influences working memory outcomes and to evaluate the impact of direct network engagement on cognitive effects.

By including the stimulation order variable, the investigators will adjust for the possibility that subjects performance will decline over time (due to fatigue) irrespective of the stimulation condition. Supplementary analysis will assess for motor performance during each stimulation condition, with the hypothesis that high frequency stimulation will have a reduction in motor scores compared to low frequency stimulation. Post-hoc analysis will also be performed to assess the relationship between task performance and functional and structural connectivity between the STN and associative networks, assuming there is some variability in individual connectivity strengths.

ELIGIBILITY:
Inclusion Criteria:

* Those with STN DBS devices
* Those with pre- and post-operative imaging
* Those that are at least 3 months post-operative

Exclusion Criteria:

* Those unable to complete the cognitive task (due to language barriers or dementia)
* Those with significant DBS complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in working memory performance between conditions | Immediately after task performance
  Working memory performance will be assessed through a modified Sternberg task. Subjects will undergo the task with and without stimulation. Measures the main effect of stimulation condition, with hypothesis that theta stimulation of associative STN will improve performance compared to no stimulation. Outcome measured through percent of correctly recalled sequences.

SECONDARY OUTCOMES:
Interaction effect between groups and stimulation condition | Immediately after task performance
  A secondary analysis will categorize subjects into two groups: 1) those where differential targeting of the associative and sensorimotor STN networks was achieved and 2) those where differential targeting of these networks was not possible using the imaging-based criteria previously mentioned. The linear mixed-effect model will be repeated with the addition of an interaction term between group and stimulation condition. The hypothesis is that there will be a significant interaction effect between group and stimulation condition. Specifically, the investigators expect to observe an increase in working memory performance during the theta (6 Hz) stimulation of the associative STN network condition, within the subject group where differential targeting of the associative and sensorimotor STN networks was achieved.

OTHER OUTCOMES:
Correlation between working memory performance and STN connectivity | Immediately after task performance
  Connectivity of the stimulated STN region will be calculated with structural (streamline count and strength) and functional (Pearson Correlation) MRI data. The change in working memory performance will be correlated to the connectivity metrics with a linear regression. The hypothesis is that there will be a positive correlation between working memory change and connectivity strength of the STN to associative networks (higher connectivity will be related to higher working memory performance).

CONTACTS AND LOCATIONS:
Locations (1):
- Leslie and Gordan Diamond Health Care Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No